CLINICAL TRIAL: NCT04707586
Title: The Effect of Lokal Cold Application in Nitroglycerin-Induced Headache
Brief Title: Lokal Cold Application in Nitroglycerin-Induced Headache (NIH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yasemin Kalkan Uğurlu (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Yasemin Kalkan Uğurlu, Research Assistant MScN, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9080; 7bRd8d6b (Registry Identifier: Istanbul University Cerrahpasa)
Record Dates: First submitted 2020-12-23; First posted 2021-01-13 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Headache
Keywords: Cryotherapy, Headache, Nitrates,
MeSH Terms: conditions — Headache

STUDY DESIGN:
Intervention Model Description: The quasi-experimental, two-group, pretest-posttest study
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No application will be made to patients in this group. Routine patient care will be provided. After the patients who develop pain are recorded, the application will be made with a cold application bandage.
- experimental group (Experimental): Patients in this group will be applied cold application with cold application bandage for 20 minutes as soon as the infusion begins.
  Interventions: Other: Cold Application

INTERVENTIONS:
Other: Cold Application — Created by the researcher; A bandage with 3 pieces of 13x10 cm cold gel and a cold gel container in which they are placed will be used, which can be adjusted according to the head circumference of the patient between 60-80 cm in length. The ability of the cold gel cups of the bandage to be moved on the bandage will allow comfortable cold application to the patient's bilateral frontotemporal and occipital areas at the same time. After waiting for 20 minutes in the freezer part of the refrigerator, the temperature and temperature of the gels applied and the cold application area before and after each application will be measured and recorded. An Infrared Non-Contact Food Thermometer will be used for temperature measurement of cold gel packs, and an Infrared Non-Contact Thermometer device will be used for temperature measurement of the cold application area.
  Arms: experimental group

SUMMARY:
The study was planned to evaluate the effect of local cold application on headache severity in individuals who received intravenous nitroglycerin treatment, which mostly causes headache due to its vasoditator effect. It is thought that the results to be obtained may provide evidence for the development of patient care guidelines.

DETAILED DESCRIPTION:
The study was planned to evaluate the effect of local cold application on headache severity in individuals who received intravenous nitroglycerin treatment, which mostly causes headache due to its vasoditator effect.

Inclusion criteria;

* The patient's volunteerism to participate in the research,
* Over the age of 18,
* Being conscious,
* Any analgesic, NSAID, triptan etc. Not taking antimigren drugs or opioids,
* No cold allergies. Exclusion Criteria;
* Difficulty in communicating (speaking, perception, language, comprehension problems),
* Vision and / or hearing loss,
* Having a cold allergy.

Purpose and Type of Research:

This research was planned as a quasi-experimental, two-group, pretest-posttest study to determine the effect of local cold application on headache in individuals treated with intravenous NTG, which mostly causes headache due to its vasodilator effect.

Place and Time of the Study It will be carried out in Ordu State Hospital Coronary Intensive Care Unit between 15 December 2020 - 15 December November 2021.

Research Population and Sample The universe of the study is planned to be composed of all patients who were hospitalized in Ordu State Hospital Coronary Intensive Care Unit between December 2020 and December 2021 and received intravenous nitroglycerine treatment.

The sample of the study will be the patients who meet the sample selection criteria and are willing to participate in the study. The research sample will consist of experimental and control groups.

Experiment 1:Local cold application was applied to the patients with the help of the applicator during the first 20 minutes of the nitroglycerin infusion. The patient was followed up during the cold application, after the procedure, the patient was evaluated in detail using the Patient Follow-up Form and VAS, and his questions were answered. The patient was given detailed information about the application before the procedure.

Experiment 2: The patients were evaluated in detail using the Patient Follow-up Form and VAS for the first 12 hours of the infusion. Local cold application was applied for 20 minutes with the help of the applicator to the patients who developed headache. Immediately after the cold application, it was evaluated in detail using the Patient Follow-up Form and VAS. The groups were compared according to the data obtained.

Power analysis (G*Power 3.1.9.2) was performed to determine the sample size of the study. As a result of the analysis; In the evaluation made according to headache severity, the sample size determined for Power:0.80, β:0.20 and α:0.05 is a minimum of 14 patients for each group. However, to increase the reliability of the study and considering that there may be patients who could leave the study during the study, the total number of samples was determined as 70, 35 in the experimental 1 group and 35 in the experimental 2 group.

Data Collection Method

* Individuals who meet the criteria for inclusion in the sampling will be informed about the purpose, content and method of the research, and after the randomization process, experimental and control groups will be formed by obtaining the necessary written permission from those who agree to participate in the study.
* The research will consist of 2 groups as Experiment 1(Group of Local Cold Application at the Beginning of Infusion) and Experiment 2 (The Group Not Applying Local Cold at the Beginning of Infusion)
* Data will be collected by the researcher.
* Within the scope of the research, the patients in the experimental group who used the cold application bandage will be informed about the use of the bandage.
* Patient Information Form, Patient Follow-up Form and Visual Pain Perception Scale will be used to evaluate the sociodemographic, disease, treatment and pain level of all patients participating in the study prior to nitroglycerin infusion.
* A cold application bandage will be attached to the experimental 1 group and local cold application will be applied to the patient for the first 20 minutes of the nitroglycerine infusion. After 20 minutes, the bandage will be removed from the patient and the cold application will be terminated. The patient will be followed during the cold application, and the questions of the patient will be answered after the procedure. Immediately after the cold application, the patient's headache will be evaluated in detail using the Visual Pain Perception Scale and the Patient Follow-up Form.
* Patients in the experimental 2 group who develop headaches will be evaluated in detail using the Visual Pain Perception Scale and the Patient Follow-up Form, a cold application bandage will be worn and local cold application will be performed for 20 minutes. Immediately after the cold application, it will be evaluated in detail again using the Visual Pain Perception Scale and Patient Monitoring Form. In this way, the preventive and therapeutic effect of local cold application will be evaluated in patients receiving intravenous nitroglycerin treatment.
* Groups will be compared according to the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* The patient's volunteerism to participate in the research,
* Over the age of 18,
* Being conscious,
* Any analgesic, NSAID, triptan etc. Not taking antimigren drugs or opioids,
* No cold allergies.

Exclusion Criteria:

* Difficulty in communicating (speaking, perception, language, comprehension problems),
* Vision and / or hearing loss,
* Having a cold allergy.
* Blood pressure above 150/90 mm / Hg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Headache | 30 minutes, 3.,6., 9. and 12. hours after nitroglycerin infusion starts
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The distance between 'no pain' and the mark then defines the subject's pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin K Uğurlu, Principal Investigator — Ordu Üniversitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Nuray Enc, Istanbul
  - Yasemin Kalkan Uğurlu, Ordu

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be shared after the study is finished.
Supporting Information: Study Protocol
Time Frame: Data will become available towards the end of 2022 and, it can be used for 1 year.
Access Criteria: IPD Sharing will be make only for research.

REFERENCES:
- [Background] Sprouse-Blum AS, Gabriel AK, Brown JP, Yee MH. Randomized controlled trial: targeted neck cooling in the treatment of the migraine patient. Hawaii J Med Public Health. 2013 Jul;72(7):237-41. PMID 23901394
- [Background] Demir Y, Khorshid L. The effect of cold application in combination with standard analgesic administration on pain and anxiety during chest tube removal: a single-blinded, randomized, double-controlled study. Pain Manag Nurs. 2010 Sep;11(3):186-96. doi: 10.1016/j.pmn.2009.09.002. Epub 2010 May 31. PMID 20728068
- [Background] Ertug N, Ulker S. The effect of cold application on pain due to chest tube removal. J Clin Nurs. 2012 Mar;21(5-6):784-90. doi: 10.1111/j.1365-2702.2011.03955.x. Epub 2011 Nov 15. PMID 22082021
- [Result] Fraser F, Matsuzawa Y, Lee YSC, Minen M. Behavioral Treatments for Post-Traumatic Headache. Curr Pain Headache Rep. 2017 May;21(5):22. doi: 10.1007/s11916-017-0624-x. PMID 28283812
- [Result] Ucler S, Coskun O, Inan LE, Kanatli Y. Cold Therapy in Migraine Patients: Open-label, Non-controlled, Pilot Study. Evid Based Complement Alternat Med. 2006 Dec;3(4):489-93. doi: 10.1093/ecam/nel035. Epub 2006 Jun 15. PMID 17173113